CLINICAL TRIAL: NCT06694532
Title: Comparative Study Between the Effectiveness of High Versus Low Molecular Weight Hyaluronic Acid in TMJ Arthrocentesis
Brief Title: EffIcacy Between Arthrocentesis With High Versus Low Molecular Weight Hyaluronic Acid in Treatment of TMJ Disorders
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basel khaled mohamed (Other)
Responsible Party: Sponsor-Investigator, Basel khaled mohamed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyaluronic and TMJ Disorders
Record Dates: First submitted 2023-10-30; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Temporomandibular Joint Disorders; Arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Hyaluronic Acid; Arthrocentesis; Syringes

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The study will be carried out in Patients in two Groups aged between 17 to 70 years , of both sexes, who had painful symptoms, with or without presence of joint noise, and had unilateral or bilateral internal derangement of the TMJ proven by clinical examination, with no improvement after conservative treatment, were included in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high molucular weight hyalurinic acid . (Experimental): patients injected e high molucular weight hyalurinic acid .
  Interventions: Drug: Hyaluronic acid; Device: Syringes
- low molcular weight hyaurinic acid (Experimental): patients injected with low molucular weight hyalurinic acid .
  Interventions: Drug: Hyaluronic acid; Device: Syringes

INTERVENTIONS:
Drug: Hyaluronic acid — Comparative study between Hyalgan and Hyorth injectable products in TMJ Disorders by arthrocentesis of 2 syringes device
  Other Names: Arthrocentesis
Device: Syringes — Whilst you are asleep, two small needles will be inserted into the TMJ / Jaw Joint. One of these needles allows sterile saline to be pumped into the joint under pressure whilst the other needle allows the saline to drain out of the joint then injection of the HA injectiable products .
  Other Names: Arthrocentesis

SUMMARY:
The study will be carried out in Patients in two Groups aged between 17 to 70 years , of both sexes, who had painful symptoms, with or without presence of joint noise, and had unilateral or bilateral internal derangement of the TMJ proven by clinical examination, with no improvement after conservative treatment.

DETAILED DESCRIPTION:
The MEASUREMENT TOOL of the study will be carried out by 2 groups the first will be injected by high molecular weight hyaluronic acid and the second wil be injected by low molecular weight hyaluronic acid Then compare between Efectevness of injection of high-molecular weight versus Low moecular weight hyaluronic acid after two-needle arthrocentesis in improving the signs and symptoms of intra-articular TMJ disorder.

, 1- significantly improving the pain on scale 1-10 , and 2-significant improvements in mouth opening range in mm by the distance between the edges of the frontal incisors with a ruler or caliper and joint noise.

3-The presence of absence of clicking and cracking in jaw .

ELIGIBILITY:
Inclusion Criteria:

* Pain or tenderness of the jaw
* Pain in one or both of the temporomandibular joints
* Aching pain in and around your ear
* Difficulty chewing or pain while chewing
* Aching facial pain
* Locking of the joint,

Exclusion Criteria:

* Muscular TMJ disorders
* Bleeding tendency

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
EFFICACY between injection of high versus low molecular weight hyaluronic acid in TMJ arthrocentesis | 36 months
  The MEASUREMENT TOOL of the study will be carried out by 2 groups the first will be injected by high molecular weight hyaluronic acid and the second wil be injected by low molecular weight hyaluronic acid Then compare between Efectevness of injection of high-molecular weight versus Low moecular weight hyaluronic acid after two-needle arthrocentesis in improving the signs and symptoms of intra-articular TMJ disorder.
  , 1- significantly improving the pain on scale 1-10 , and

SECONDARY OUTCOMES:
comparative between injection of high versus low molecular weight hyaluronic acid in TMJ arthrocentesis | 36 months
  The MEASUREMENT TOOL of the study will be carried out by 2 groups the first will be injected by high molecular weight hyaluronic acid and the second wil be injected by low molecular weight hyaluronic acid Then compare between Efectevness of injection of high-molecular weight versus Low moecular weight hyaluronic acid after two-needle arthrocentesis in improving the signs and symptoms of intra-articular TMJ disorder.
  2-significant improvements in mouth opening range in mm by the distance between the edges of the frontal incisors with a ruler or caliper and joint noise.

CONTACTS AND LOCATIONS:
Overall Officials: Basel K Mohamed, Principal Investigator — Assiut Univeristy
Locations (1):
- Assiut Univeristy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No